CLINICAL TRIAL: NCT03249714
Title: A 24-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Ofatumumab in Patients With Relapsing Multiple Sclerosis Followed by an Extended Treatment of at Least 24 Weeks With Open-label Ofatumumab
Brief Title: Efficacy and Safety of Ofatumumab Compared to Placebo in Patients With Relapsing Multiple Sclerosis Followed by Extended Treatment With Open-label Ofatumumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMB157G1301
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: double-blind; placebo controlled; ofatumumab; relapsing multiple sclerosis; Japanese patients; MS; RMS; adult; OMB157
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMB 20 mg (Experimental): Ofatumumab 20 mg subcutaneous injection on Days 1,7, 14 and every 4 weeks for 24 weeks in Core. Core placebo patients received loading dose at Weeks 25 and 26 and then all Extension patients received dose every 4 Weeks up to Week 48.
  Interventions: Drug: Ofatumumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection matching to ofatumumab every 4 weeks for 24 weeks in Core
  Interventions: Drug: Matching placebo of ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Provided in pre-filled syringes for subcutaneous injection (s.c.) administration containing 20 mg ofatumumab (50 mg/mL, 0.4 mL content)
  Arms: OMB 20 mg
Drug: Matching placebo of ofatumumab — Matching placebo in pre-filled syringes
  Arms: Placebo

SUMMARY:
The study provided efficacy, safety, and pharmacokinetics (PK) data for patients with relapsing multiple sclerosis (RMS) in Japan and the other countries

DETAILED DESCRIPTION:
This study had 2 parts: A controlled Core and an open-label Extension.

* Core part: A 24-week, randomized, double-blind, placebo controlled, parallel-group, multicenter study evaluated the efficacy, safety and tolerability and PK of ofatumumab in patients with RMS.
* Extension part: The Core part was followed by an Extension part in which all patients received open-label ofatumumab. In the Extension part, patients were treated for at least 24 weeks and no longer than 48 weeks.

Sixty-four patients were randomized in a 2:1 ratio to ofatumumab or placebo in the Core part; half of the study patients were from Japan and the other half from the other countries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (MS)
* Relapsing MS (RMS)
* At least 1 appearance of a new neurological abnormality or worsening of pre-existing neurological abnormality during the previous 2 years prior to Screening AND an MRI activity (Gd-enhancing T1 lesions or new or enlarging T2 lesions) in brain during the previous 1 year prior to randomization
* EDSS score of 0 to 5.5

Exclusion Criteria:

* Primary progressive MS or SPMS without disease activity
* Patients with an active chronic disease of the immune system other than MS
* Patients at risk of developing or having reactivation of hepatitis
* Patients with active systemic infections or with neurological findings consistent with PML

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (11):
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
- Russia (2):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Novosibirsk

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=969

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients where randomized in a 2:1 ratio to ofatumumab or placebo in the Core Part
Groups:
- OMB 20 mg: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections every 4 weeks
- Placebo - OMB 20 mg: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections at Week 24, Week 25, Week 26 and every 4 weeks thereafter
Period: Double-blind Treatment (Core Part)
Arm/Group | OMB 20 mg | Placebo - OMB 20 mg
Started | 43 | 21
Completed | 40 | 19
Not Completed | 3 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Subject/guardian decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Open-label Treatment (Extension Part)
Arm/Group | OMB 20 mg | Placebo - OMB 20 mg
Started | 40 | 19
Completed | 38 | 19
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections at Week 24, Week 25, Week 26 and every 4 weeks thereafter
- Total: Total of all reporting groups
Arm/Group | OMB 20 mg | Placebo | Total
Number analyzed (Participants) | 43 | 21 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (9.49) | 35.5 (8.93) | 35.2 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 19 | 55
  Male | 7 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 21 | 11 | 32
  White | 22 | 10 | 32
Country of Enrollment [Count of Participants; unit: Participants]
  Japan | 21 | 11 | 32
  Russia | 22 | 10 | 32
Number of relapses in the past 12 months prior to screening [Mean (Standard Deviation); unit: Number of relapses] — Reported numbers are from investigator records.
  Number of relapses | 1.6 (0.90) | 1.2 (0.70) | 1.5 (0.85)
Number of Gd-enhancing T1 lesions [Mean (Standard Deviation); unit: lesions] — Magnetic Resonance Imaging (MRI) scans of the brain were were read by the central MRI reading center. The central reading center was blinded with no access to information on treatment assignments Population: n=number of participants with non-missing values
  lesions
    number analyzed (Participants) | 42 | 21 | 63
    (all) | 1.3 (2.62) | 1.0 (1.47) | 1.2 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Gadolinium-enhancing T1 Lesions Per MRI Scan - Core Part
Description: Total number of Gd-enhancing T1 lesions across scans at Week 12, 16, 20, and 24 were adjusted for the different numbers of scans. This was calculated as a rate for population, rather than at patient level, using a negative binomial regression model with log link. The model included each patient's total number of Gd-enhancing T1 lesions as the response variable, and treatment, region, and subgroup of baseline number of Gd-enhancing T1 lesions (0 or >=1) as explanatory variables, and logarithm of the patient's number of scans as the offset variable.
Time Frame: Baseline up to Week 24
Population: Full analysis set (participants with missing baseline or post-baseline MRI data could not be included in the analysis)
Measure: Number (95% Confidence Interval); unit: lesions per scan
Groups:
- OMB 20 mg: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter.
- Placebo: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter.
Arm/Group | OMB 20 mg | Placebo
Number analyzed (Participants) | 39 | 20
lesions per scan | 0.0670 [0.027 to 0.167] | 1.0413 [0.465 to 2.331]
Statistical Analysis 1: Comparison: OMB 20 mg vs Placebo; Test type: Superiority; p < 0.001, negative binominal regression model; Rate ratio = 0.064, 95% CI 2-sided [0.018 to 0.232]

2. Secondary Outcome: Number of Gadolinium-enhancing T1 Lesions Per MRI Scan - Japan vs Non-Japan - Core Part
Description: Total number of Gd-enhancing T1 lesions across scans at Week 12, 16, 20, and 24 were adjusted for the different numbers of scans. This was calculated as a rate for population, rather than at patient level, using a negative binomial regression model with log link. The model included each patient's total number of Gd-enhancing T1 lesions as the response variable, and treatment, region, subgroup of baseline number of Gd-enhancing T1 lesions (0 or >=1), and the treatment-by-region interaction term as explanatory variables, and the patient's number of scans as the offset variable.
Time Frame: Baseline up to Week 24
Population: Full analysis set (participants with missing baseline or post-baseline MRI data could not be included in the analysis)
Measure: Number (95% Confidence Interval); unit: lesions per scan
Groups:
- OMB 20 mg Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter - Japanese patients
- Placebo Japan: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter - Japanese patients
- OMB 20 mg Non-Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter
  - non-Japanese patients
- Placebo Non-Japan: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter - non-Japanese patients
Arm/Group | OMB 20 mg Japan | Placebo Japan | OMB 20 mg Non-Japan | Placebo Non-Japan
Number analyzed (Participants) | 19 | 10 | 20 | 10
lesions per scan | 0.1999 [0.082 to 0.485] | 1.4682 [0.538 to 4.004] | 0.0000 [0.0000 to 0.0000] | 0.6774 [0.234 to 1.962]
Statistical Analysis 1: Comparison: OMB 20 mg Japan vs Placebo Japan; Test type: Superiority; p = 0.003, negative binomial regression — Statistical significance (2-sided) at the 0.05 level; rate ratio = 0.136, 95% CI 2-sided [0.036 to 0.513]
Statistical Analysis 2: Comparison: OMB 20 mg Non-Japan vs Placebo Non-Japan; Test type: Superiority; p < 0.001, negative binominal regression; Indicates statistical significance (2-sided) at the 0.05 level; rate ratio = 0.000, 95% CI 2-sided [0.000 to 0.000]

3. Secondary Outcome: Number of New or Enlarging T2 Lesions on MRI Scans (Annualized T2 Lesion Rate) - Core Part
Description: Number of new/enlarging T2 lesions on the last available MRI scan in the Core Part (up to Week 24) relative to baseline, adjusted for different follow-up times. This was calculated as a rate for population, rather than at patient level, using a negative binomial regression model with log-link. The model included each patient's last available number of new or enlarging T2 lesions relative to baseline as the response variable, and treatment, region, subgroup of baseline number of Gd-enhancing T1 lesions (0 or >=1), and baseline volume of T2 lesions as explanatory variables, and the patient's follow-up time as the offset variable.
Time Frame: Baseline up to Week 24
Population: Full analysis set (participants with missing baseline or post-baseline MRI data could not be included in the analysis)
Measure: Number (95% Confidence Interval); unit: T2 lesions per year
Arm/Group | OMB 20 mg | Placebo
Number analyzed (Participants) | 40 | 20
T2 lesions per year | 3.7344 [2.354 to 5.925] | 13.1533 [7.197 to 24.039]
Statistical Analysis 1: Comparison: OMB 20 mg vs Placebo; Test type: Superiority; p = 0.002, negative binominal regression; Rate ratio = 0.284, 95% CI 2-sided [0.130 to 0.620]

4. Secondary Outcome: Annualized Relapse Rate (ARR) - Core Part
Description: ARR was the number of confirmed MS relapses in a year. A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system). ARR was calculated as a rate for population, rather than at patient-level, using a negative binomial regression model with log-link. The model included each patient's number of confirmed relapses as the response variable, and treatment and region as explanatory variables, and the patient's follow-up time as the offset variable.
Time Frame: Baseline up to Week 24
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: relapses in a year
Arm/Group | OMB 20 mg | Placebo
Number analyzed (Participants) | 43 | 21
relapses in a year | 0.2640 [0.111 to 0.629] | 0.6286 [0.276 to 1.430]
Statistical Analysis 1: Comparison: OMB 20 mg vs Placebo; Test type: Superiority; p = 0.119, negative binominal regression; Rate ratio = 0.420, 95% CI 2-sided [0.141 to 1.250]

5. Secondary Outcome: Pharmacokinetic (PK) Concentrations of Ofatumumab - Core Part
Description: Blood samples were collected at the scheduled visit. Summary statistics of PK concentrations from trough samples.
Time Frame: Pre-dose at Baseline, Days 2, 5, 7, 14, Weeks 4, 12, 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- OMB 20 mg Non-Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter - non - Japanese patients
- OMB 20 mg - All Patients: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter
Arm/Group | OMB 20 mg Japan | OMB 20 mg Non-Japan | OMB 20 mg - All Patients
Number analyzed (Participants) | 21 | 22 | 43
ug/mL
  Baseline n=21,22,43 | 0.03 (0.07) | 0.9 (.39) | .06 (.28)
  Day 2 n=21,22,43 | .43 (.38) | .24 (.32) | 0.33 (.36)
  Day 5 n=21,22,43 | .88 (.40) | .60 (.46) | .73 (.45)
  Day 7 n=21,22,43 | .84 (.39) | 0.48 (.34) | 0.66 (.40)
  Day 14 n=21,22,43 | 2.17 (.63) | 1.71 (1.00) | 1.93 (.86)
  Week 4 n=21,22,43 | 2.69 (.86) | 2.03 (1.14) | 2.35 (1.05)
  Week 12 n=20,21,41: number analyzed (Participants) | 20 | 21 | 41
  Week 12 n=20,21,41 | .66 (.62) | 0.38 (.38) | .51 (.53)
  Week 24 n=20,20,40: number analyzed (Participants) | 20 | 20 | 40
  Week 24 n=20,20,40 | .84 (.60) | .64 (.46) | .74 (.54)

6. Secondary Outcome: B-cell Counts - Japan vs Non-Japan - Core Part
Description: Blood samples were collected at the scheduled visits. The CD19+ B-cell counts were measured by the central laboratory.
Time Frame: Baseline, Days 2, 5, 7, 14, Weeks 4, 12, 24
Population: Safety set
Measure: Median (Full Range); unit: cells/uL
Groups:
- OMB 20 mg Non-Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter- non-Japanese participants
Arm/Group | OMB 20 mg Japan | Placebo Japan | OMB 20 mg Non-Japan | Placebo Non-Japan
Number analyzed (Participants) | 21 | 11 | 22 | 10
cells/uL
  Baseline n=21,11,22,9: number analyzed (Participants) | 21 | 11 | 22 | 9
  Baseline n=21,11,22,9 | 207 [41 to 566] | 205 [81 to 814] | 208 [78 to 419] | 244 [81 to 385]
  Day 2 n=21,11,21,9: number analyzed (Participants) | 21 | 11 | 21 | 9
  Day 2 n=21,11,21,9 | 3.0 [1 to 69] | 319.0 [127 to 629] | 14.0 [1 to 283] | 292.0 [79 to 797]
  Day 5 n=20,10,14,7: number analyzed (Participants) | 20 | 10 | 14 | 7
  Day 5 n=20,10,14,7 | 3.0 [1 to 50] | 216.5 [91 to 658] | 8.5 [0 to 300] | 257.0 [124 to 533]
  Day 7 n=21,11,22,9: number analyzed (Participants) | 21 | 11 | 22 | 9
  Day 7 n=21,11,22,9 | 3.0 [0 to 21] | 209.0 [61 to 514] | 3.5 [0 to 37] | 228.0 [15 to 319]
  Day 14 n=21,11,19,8: number analyzed (Participants) | 21 | 11 | 19 | 8
  Day 14 n=21,11,19,8 | 2 [0 to 24] | 266.0 [82 to 496] | 3.0 [0 to 19] | 226.0 [132 to 323]
  Week 4 n=21,10,21,8: number analyzed (Participants) | 21 | 10 | 21 | 8
  Week 4 n=21,10,21,8 | 1.0 [0 to 19] | 235.5 [178 to 489] | 1.0 [0 to 7] | 179.5 [15 to 353]
  Week 12 n=20,10,18,9: number analyzed (Participants) | 20 | 10 | 18 | 9
  Week 12 n=20,10,18,9 | 1.0 [0 to 8] | 211.0 [130 to 464] | 1.0 [0 to 8] | 200.0 [59 to 316]
  Week 24 n=19,8,19,8: number analyzed (Participants) | 19 | 8 | 19 | 8
  Week 24 n=19,8,19,8 | 0.0 [0 to 4] | 227.5 [79 to 462] | 1.0 [0 to 15] | 224.5 [106 to 523]

7. Secondary Outcome: Number of Gadolinium-enhancing T1 Lesions Per MRI Scan - Extension Part
Description: Total number of Gd-enhancing T1 lesions per scan during the Extension Part (up to Week 48) calculated as a rate for population, rather than at patient-level. It was calculated as sum of each patient's total number of Gd-enhancing T1 lesions across scans at Week 36 and 48, divided by sum of each patient's total number of scans.
Time Frame: Week 24 up to Week 48
Population: Extension full analysis set
Measure: Number; unit: lesions per scan
Groups:
- Placebo (Core) - OMB 20 mg (Extension): CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections at Week 24, Week 25, Week 26 and every 4 weeks thereafter
Arm/Group | OMB 20 mg | Placebo (Core) - OMB 20 mg (Extension)
Number analyzed (Participants) | 38 | 19
lesions per scan | 0.027 | 0.025

8. Secondary Outcome: Number of New or Enlarging T2 Lesions on MRI Scans (Annualized T2 Lesion Rate) - Extension Part
Description: Number of new/enlarging T2 lesions on the last available MRI scan in the Extension Part (up to Week 48) relative to Week 24, adjusted for different follow-up times. Annualized rate of new or enlarging T2 lesions was calculated by dividing the sum of each patient's number of new or enlarging T2 lesions relative to Week 24 by the sum of each patient's number of MRI assessment days during the Extension part, and then multiplying it by 365.25.
Time Frame: Week 24 up to Week 48
Population: Extension full analysis set
Measure: Number; unit: T2 lesions per year
Arm/Group | OMB 20 mg | Placebo (Core) - OMB 20 mg (Extension)
Number analyzed (Participants) | 40 | 19
T2 lesions per year | 0.230 | 0.813

9. Secondary Outcome: Annualized Relapse Rate (ARR) - Extension Part
Description: ARR was the number of confirmed MS relapses in a year. A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system). ARR (time-based) was calculated by summing each patient's number of confirmed relapses observed during the Extension part, divided by the total number of each patient's days in a study of all patients during the Extension part, and multiplied by 365.25.
Time Frame: Week 24 up to Week 48
Population: Extension full analysis set
Measure: Number; unit: relapses in a year
Arm/Group | OMB 20 mg | Placebo (Core) - OMB 20 mg (Extension)
Number analyzed (Participants) | 40 | 19
relapses in a year | 0.081 | 0.083

10. Secondary Outcome: Pharmacokinetic (PK) Concentrations of Ofatumumab - Extension Part
Description: Blood samples were collected at the scheduled visits. Summary statistics of PK concentrations from trough samples.
Time Frame: Weeks 24, 28, 36, 48
Population: Extension full analysis set
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- OMB 20 mg Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections every 4 weeks - Japanese patients
- OMB 20 mg Non-Japan: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections every 4 weeks - non-Japanese patients
Arm/Group | OMB 20 mg Japan | OMB 20 mg Non-Japan
Number analyzed (Participants) | 20 | 20
ug/mL
  Week 24 | .84 (.60) | .64 (.46)
  Week 28 n=19,19: number analyzed (Participants) | 19 | 19
  Week 28 n=19,19 | 0.64 (.36) | .61 (.48)
  Week 36 n=19,19: number analyzed (Participants) | 19 | 19
  Week 36 n=19,19 | .97 (.53) | .72 (.56)
  Week 48 n=18,19: number analyzed (Participants) | 18 | 19
  Week 48 n=18,19 | 1.11 (.56) | .94 (.76)

11. Secondary Outcome: B-cell Counts - Extension Part
Description: Blood samples were collected at the scheduled visits. The CD19+ B-cell counts were measured by the central laboratory.
Time Frame: Weeks 24, 36 and 48
Population: Extension safety set
Measure: Median (Full Range); unit: cells/uL
Arm/Group | OMB 20 mg | Placebo (Core) - OMB 20 mg (Extension)
Number analyzed (Participants) | 40 | 19
cells/uL
  Week 24 n=40,18: number analyzed (Participants) | 40 | 18
  Week 24 n=40,18 | 0.0 [0 to 15] | 1.0 [0 to 5]
  Week 36 n=38, 9: number analyzed (Participants) | 38 | 9
  Week 36 n=38, 9 | 0.5 [0 to 4] | 1.0 [0 to 2]
  Week 48 n=38,1: number analyzed (Participants) | 38 | 1
  Week 48 n=38,1 | 1.0 [0 to 4] | 4.0 [4 to 4]

12. Secondary Outcome: Participants With Confirmed Relapse - Core and Extension Parts
Description: A confirmed MS relapse was defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system).
Time Frame: Baseline up to Week 48
Population: Extension full analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Core) - OMB 20mg (Extension): CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter. EXTENSION PART: Ofatumumab 20 mg s.c. injections at Week 24, Week 25, Week 26 and every 4 weeks thereafter
Arm/Group | OMB 20 mg | Placebo (Core) - OMB 20mg (Extension)
Number analyzed (Participants) | 40 | 19
Participants
  Day 1 to Week 12 | 3 | 2
  >Week 12 to Week 24 | 1 | 4
  >Week 24 to Week 36 | 1 | 0
  >Week 36 to Week 48 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until last administration of study treatment plus 100 days post treatment, up to maximum duration of approximately 638 days
Groups:
- OMB 20mg Core: CORE PART: Ofatumumab 20 mg s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter
- Placebo Core: CORE PART: Placebo s.c. injections on Days 1, 7, 14, Week 4 and every 4 weeks thereafter
- OMB 20mg Continued: EXTENSION PART: Ofatumumab 20 mg s.c. injections every 4 weeks
- OMB 20mg Switched (From Placebo): EXTENSION PART: Ofatumumab 20 mg s.c. injections at Week 24, Week 25, Week 26 and every 4 weeks thereafter
Arm/Group | OMB 20mg Core | Placebo Core | OMB 20mg Continued | OMB 20mg Switched (From Placebo)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/21 | 0/40 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/21 | 1/40 | 0/19
Other Adverse Events (participants affected / at risk) | 23/43 | 15/21 | 23/40 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg Core (N=43) | Placebo Core (N=21) | OMB 20mg Continued (N=40) | OMB 20mg Switched (From Placebo) (N=19)
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMB 20mg Core (N=43) | Placebo Core (N=21) | OMB 20mg Continued (N=40) | OMB 20mg Switched (From Placebo) (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 1 | 2 | 2 | 1
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 4 | 7 | 4
Oral herpes (Infections and infestations) | 4 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 1 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 9 | 4 | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 1
Tension headache (Nervous system disorders) | 4 | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT03249714/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT03249714/SAP_001.pdf